CLINICAL TRIAL: NCT02095288
Title: Broad-spectrum Lipidomics Screening of Anti-inflammatory Drugs and Drug Candidates in In Vitro Human Whole-blood Assay (hWBA)
Brief Title: Lipidomics Screening of Anti-inflammatory Drugs and Drug Candidates in Vitro - Part A
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 818658
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: lipidomics; in vitro human whole blood assay; anti-inflammatory drugs; Lipidomics screening of anti-inflammatory drugs
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Thirty (n=30) healthy, non-smoking male and female volunteers between the ages of 18-50 will be included in this study. If all inclusion/exclusion criteria are met, a blood collection of 104 ml will be obtained and the study visit will be completed. If eligible, a volunteer may participate in this study up to four separate times, but not more than two times in the same week.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers: Blood draw
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — This is a single blood donation, no drugs or devices administered
  Other Names: It's a single blood draw of 104 ml in total

SUMMARY:
Cardiovascular complications of NSAIDs, selective for inhibition of COX-2, stimulated interest in microsomal prostaglandin E synthase-1 (mPGES-1) as an alternative drug target. Global deletion of mPGES-1 in mice suppresses PGE2 and augments PGI2 by PGH2 substrate rediversion. Unlike COX-2 inhibition or gene deletion, mPGES-1 deletion does not cause a predisposition to thrombogenesis and hypertension. However, cell-specific deletion of mPGES-1 reveals that the predominant substrate rediversion product amongst the prostaglandins varies by cell type, complicating drug development. We have developed an ultra performance liquid chromatography/ tandem mass spectrometry (UPLC-MS/MS) technique that allows the quantification of a wide range of lipids beyond the prostaglandin pathway (leukotrienes, anandamide and the 2-arachidonylglycerol cascades).

This study is designed to examine different pathway interventions from the arachidonic acid cascade by anti-inflammatory compounds (with a focus on mPGES-1 inhibition) in whole human blood in vitro (Part A) and ex vivo (Part B). In Part A, whole human blood will be donated by healthy volunteers and treated with screening compounds in vitro (outside of the body). Experiments will be performed to measure an array of lipids in plasma and serum from pre-stimulated whole blood treated with a single or a combination of the test compounds.

This study may reveal pathways previously unknown to be affected by the existing anti-inflammatory drugs and drug candidates, and will possibly suggest new indications and/or side effects.

DETAILED DESCRIPTION:
Nonsteroidal anti-inflammatory drugs (NSAIDs), selective for inhibition of cyclooxygenase (COX)-2, alleviate pain and inflammation by suppressing COX-2-derived prostacyclin (PGI2) and prostaglandin (PG) E2 (1). However, eight placebo-controlled clinical trials have revealed that NSAIDs, designed to inhibit specifically COX-2, predispose patients to increased cardiovascular risks including myocardial infarction, stroke, systemic and pulmonary hypertension, congestive heart failure, and sudden cardiac death (1-3). The cardiovascular adverse effects are attributable to the suppression of COX-2-derived PGI2, a potent vasodilator and inhibitor of platelet activation (4; 5). Our laboratory has shown that global deletion, selective inhibition or mutation of COX-2, or deletion of the receptor for PGI2 elevate blood pressure and accelerate thrombogenesis in mouse models (6). We have further demonstrated that vascular COX-2 deletion predisposes mice to thrombosis and hypertension (7), and that selective deletion of COX-2 in cardiomyocytes leads to cardiac dysfunction and enhanced susceptibility to induced arrhythmogenesis (8) that may contribute to the heart failure and cardiac arrhythmias reported in patients taking NSAIDs specific for inhibition of COX-2.

This cardiovascular hazard from NSAIDs prompted interest in the microsomal prostaglandin E synthase-1 (mPGES-1) as an alternative drug target. mPGES-1 is the inducible PG terminal synthase that acts downstream of COX-2 and catalyzes the conversion of the intermediate COX endoperoxide product PGH2 to PGE2 (9). We have previously reported that similar to the interference with COX-2 expression or function, global or cell-specific deletion of mPGES-1 suppresses PGE2 production; but unlike with COX-2, global mPGES-1 deficiency augments biosynthesis of PGI2 and does not predispose normo- or hyperlipidemic mice to thrombogenic or hypertensive events (9-11). Both suppression of PGE2 and augmentation of PGI2 in mPGES-1-/- mice result from the rediversion of the accumulated PGH2 substrate to PGI2 synthase (10). Furthermore, global deletion of mPGES-1 limits the vascular proliferative response to wire injury (12), retards atherogenesis and suppresses angiotensin II-induced abdominal aortic aneurysm formation in hyperlipidemic mice (10; 13). We have also shown that mPGES-1-deficiency does not affect ozone-induced airway inflammation or airway hyper-responsiveness suggesting that pharmacological inhibition of mPGES-1 and endoperoxide rediversion to PGD2 may not predispose patients at risk to airway dysfunction (14). In addition, studies by others indicate that global deletion of mPGES-1 reduces the post-ischemic brain infarction and neurological dysfunction in cerebral ischemia/reperfusion in mice (15). mPGES-1 deficiency also renders mice less susceptible to excessive inflammation and hypersensitivity in rodent models of analgesia (16; 17). Taken together, these findings suggest that pharmacological inhibition of mPGES-1 may retain anti-inflammatory effects from PGE2 suppression, but due to PGI2 augmentation, targeting of mPGES-1 might avoid the cardiovascular risks associated with selective COX-2 inhibitors.

PGH2 substrate rediversion consequent to mPGES-1 deletion is a ubiquitous event observed at the cellular level and systemically (urinary prostaglandin metabolites); the profile of the rediversion products, however, varies by cell and tissue type, the disease model, and the extent of system perturbation (6; 10-14; 18-21). We have shown that in mice deficient in mPGES-1 in endothelial cells (EC) or vascular smooth muscle cells (VSMC), PGI2 is the predominant substrate rediversion product, whereas deletion of mPGES-1 in myeloid cells results in shunting of PGH2 mostly towards TxA2(11). Functionally, mice lacking mPGES-1 in myeloid cells, exhibited a poor response to vascular injury implicating myeloid mPGES-1 as a cardiovascular drug target. Therefore, cell-specific mPGES-1 deletion leads to a differential pattern of substrate rediversion and may affect biological function of the system, thus complicating drug development. What is unknown is whether genetic deletion or pharmacological inhibition of mPGES-1 can directly (through substrate rediversion) or indirectly (by effects of prostaglandin rediversion products on enzyme expression or their further metabolism to transcellular products (22)) influence the lipidome beyond the prostaglandin pathway with functional consequence. For example, disruption of AA-PGE2 metabolism might influence arachidonate product formation by the cytochrome P450 (23; 24), leukotriene, anandamide, 2-arachidonylglycerol (2-AG) and other cascades (25). At the cellular level, mPGES-1-/- macrophages, pretreated with LPS and stimulated with arachidonic acid (AA), exhibit a 5-fold increase in 12-HHT (12-hydroxyheptadecatrienoic acid), indicating substrate rediversion towards thromboxane A synthase (18). Inhibition and deletion of COX-2 have been reported to augment metabolites of 5-lipoxygenase (5-LO) pathway 5-HETE (5-hydroxyeicosatetraenoic acid) and leukotrienes LTB4, LTC4, LTD4 (26-28), and metabolites of CYP450 cascade 14,15-DHET/EET (dihydroxyeicosatrienoic/epoxyeicosatrienoic acid) (26). Therefore, the substrate AA may be shunted from one pathway to the other when a particular branch of the cascade is pharmacologically inhibited or genetically ablated.

Here, we will conduct a broad-spectrum lipidomics screening of anti-inflammatory drugs and drug candidates that antagonize receptors (LTC4, LTB4, EP4 receptors) or inhibit specific components (COX-1, COX-2, mPGES-1, 5-KO, FLAP, LTA4A) of arachidonic acid pathway in an in vitro human whole-blood assay (hWBA). Healthy, non-smoking, male and female volunteers will be asked to donate blood. Human whole blood assays will include (i) determination of the baseline lipid levels at various time points in stimulated whole blood, (ii) measurement of lipids in pre-stimulated whole blood treated with a single intervention compound, (iii) quantitation of lipids in pre-stimulated whole blood treated with a combination of intervention compounds. We expect that the compounds at focus will affect various inflammatory pathways resulting in new patterns of substrate rediversion and measurement of previously unknown lipid products.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-50
* non-pregnant females
* non-smoking males and females
* in good health as based on medical history

Exclusion Criteria:

* Subjects with any medical condition, which according to the investigator, may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject.
* Subjects who have received an experimental drug within 30 days prior to the study
* Subjects who have taken medications at least two weeks prior to the study. Subjects using hormonal birth control, however, will not be an exclusionary criterion.
* Subjects who have taken aspirin or aspirin containing products for at least two weeks prior to the study.
* Subjects who have taken acetaminophen, NSAIDs, COX-2 inhibitors (OTC or prescription) for at least two weeks prior to the study.
* Subjects who are consuming any type of tobacco product(s).
* Subjects who consume high doses of antioxidant vitamins daily (vitamin C> 1000mg, Vitamin E> 400IU, Beta Carotene> 1000IU, Vitamin A> 5000IU, Selenium> 200mcg, Folic Acid> 1mg) for the two weeks prior to the start of the study and throughout the study.
* Subjects who consume alcohol, caffeine or high fat food 24 hours prior to the study.

  * Pregnant female subjects

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal, healthy, non-smoking, male and non-pregnant female volunteers between the ages of 18 - 50
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Quantification of lipids in plasma and serum from the whole blood treated with the test compounds | Within a week after the blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Garret A FitzGerald, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- The Clinical Translational Research Center (CTRC) at the Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mazaleuskaya LL, Salamatipour A, Sarantopoulou D, Weng L, FitzGerald GA, Blair IA, Mesaros C. Analysis of HETEs in human whole blood by chiral UHPLC-ECAPCI/HRMS. J Lipid Res. 2018 Mar;59(3):564-575. doi: 10.1194/jlr.D081414. Epub 2018 Jan 4. PMID 29301865